CLINICAL TRIAL: NCT05805852
Title: Challenges in Management of Abdominal Trauma in Sohag University Hospital A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maikel Ashraf Sabry, micheal ashraf sabry, Sohag University
Other Study IDs: Soh-Med-23-03-13MS
Record Dates: First submitted 2023-03-17; First posted 2023-04-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Abdominal Trauma
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with surgical intervention
- patients with no surgical intervention

SUMMARY:
The present study will be conducted to evaluate the different patterns of abdominal trauma patients and their management in the Emergency Department of Sohag University Hospital

DETAILED DESCRIPTION:
The present study will be conducted to evaluate the different patterns of abdominal trauma patients and their management in the Emergency Department of Sohag University Hospital This study will be a prospective study which will be conducted at the Emergency Department of Sohag University Hospital the study population include all patients with abdominal trauma

ELIGIBILITY:
Inclusion Criteria:

* any patient presented with abdominal trauma

Exclusion Criteria:

* Patients with extra abdominal injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any patient presented with abdominal trauma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
mortality at final follow up | one month

SECONDARY OUTCOMES:
morbidity | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No